CLINICAL TRIAL: NCT00814801
Title: Placebo-controlled Confirmatory Study of Galantamine (R113675) for Alzheimer's Type Dementia
Brief Title: An Efficacy and Safety Study of Galantamine for the Treatment of Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR010297; GAL-JPN-5 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Cognitive dysfunction; Dementia; Galantamine; R113675
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Galantamine 16 mg/day (Experimental)
  Interventions: Drug: Galantamine 16 mg/day
- Galantamine 24 mg/day (Experimental)
  Interventions: Drug: Galantamine 24 mg/day

INTERVENTIONS:
Drug: Placebo — Form= tablet, route= oral use. Corresponding placebo tablets confirmed to be indistinguishable from the galantamine tablets will be administered for 24 weeks.
  Arms: Placebo
Drug: Galantamine 16 mg/day — Type= exact number, number= 8, 16, unit= mg/day, form= tablet, route= oral use. Patients will receive 8 mg galantamine daily for the first 4 weeks, and 16 mg galantamine daily for the remaining 20 weeks.
  Arms: Galantamine 16 mg/day
Drug: Galantamine 24 mg/day — Type= exact number, number= 8, 16, 24, unit= mg/day, form= tablet, route= oral use. Patients will receive 8 mg galantamine daily for the first 4 weeks, then 16 mg galantamine daily for the following 4 weeks, and 24 mg galantamine daily for the remaining 16 weeks.
  Arms: Galantamine 24 mg/day

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two fixed doses (16mg/day and 24mg/day) of galantamine (a drug for treating dementia) versus placebo for the treatment of patients with Alzheimer's disease.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither the physician nor the patient know the name of the study medication), placebo-controlled, parallel-group study to evaluate the efficacy and safety of two fixed doses of galantamine (16 and 24 milligrams per day [mg/day]) in patients with Alzheimer's disease. The study consists of a 4-week screening period during which all patients will receive placebo, and a 24-week double-blind treatment period during which patients will receive placebo, galantamine 16 mg/day, or galantamine 24 mg/day. For patients receiving galantamine treatment, the starting dose is 8 mg/day and increases at 4-week intervals in increments of 8 mg/day. The primary measures of effectiveness are the change from baseline to the end of the study (week 24) in the Alzheimer's Disease Assessment Scale - Japan cognitive subscale (ADAS-J cog) and the Clinician's Interview-Based Impression of Change plus - Japan (CIBIC plus-J). Safety assessments include the incidence of adverse events, clinical laboratory tests, vital signs, electrocardiograms (ECGs), and physical examination findings. The study hypothesis is that galantamine will be effective in the treatment of Alzheimer's disease. Study drug taken orally twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of Alzheimer's disease according to the National Institute of Neurological and Communicative Disorders and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* Having a Mini-Mental Status Examination (MMSE) score of 10 - 22 inclusive
* Having an Alzheimer's Disease Assessment Scale - Japan cognitive subscale (ADAS-J cog) score of at least 18
* Exhibiting an onset and progression of cognitive dysfunction during at least 6 months prior to the screening period

Exclusion Criteria:

* Patients with neurodegenerative diseases other than Alzheimer's disease, such as Lewy bodies disease, (dementia due to tiny round structures made of proteins that develop within nerve cells in the brain), Parkinsonism, etc
* Patients with cognitive dysfunction due to cerebral damage resulting from a lack of oxygen, a brain injury, etc
* Patients with multi-infarct dementia (brought on by a series of strokes) or active cerebrovascular disease
* Patients with clinically significant cardiovascular disease
* Patients currently taking drugs such as a cholinesterase inhibitors, which improve cerebral circulation/metabolism

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Fukuoka, Japan

REFERENCES:
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- See also: An Efficacy and Safety Study of Galantamine for the Treatment of Patients with Alzheimer's Disease. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=411&filename=CR010297_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Galantamine Group 1: Galantamine 16 mg/day
- Galantamine Group 2: Galantamine 24 mg/day
Period: Overall Study
Arm/Group | Placebo Group | Galantamine Group 1 | Galantamine Group 2
Started | 194 | 192 | 194
Completed | 160 | 154 | 151
Not Completed | 34 | 38 | 43
Not completed — Adverse Event | 15 | 16 | 19
Not completed — Withdrawal by Subject | 9 | 11 | 14
Not completed — Inappropriate as a subject | 1 | 1 | 1
Not completed — Change of patients for CIBIC plus-J | 1 | 1 | 0
Not completed — Missing or change of caregiver | 6 | 2 | 4
Not completed — Non-compliance | 0 | 1 | 1
Not completed — Other | 2 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Galantamine Group 1 | Galantamine Group 2 | Total
Number analyzed (Participants) | 191 | 191 | 192 | 574
Age, Continuous [Mean (Standard Deviation); unit: years] — Six participants were excluded from the randomized patients as no evaluation on both ADAS and CIBIC was made after treatment with study medication.
  years | 75.5 (7.6) | 75.6 (8.4) | 74.6 (8.8) | 75.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Six participants were excluded from the randomized patients as no evaluation on both Alzheimer's disease assessment scale (ADAS) and Clinician's Interview-Based Impression of Change (CIBIC) was made after treatment with study medication.
  Participants
    Female | 132 | 125 | 145 | 402
    Male | 59 | 66 | 47 | 172

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Alzheimer's Disease Assessment Scale - Japan Cognitive Subscale (ADAS-J Cog)
Description: ADAS-J cog is the Japanese version of the cognitive function subscale of the Alzheimer's disease assessment scale (ADAS). This scale is used to detect changes in cognitive function in individuals with Alzheimer disease on the basis of three domains: memory, language and behavior. The minimum score is zero (0) and means well cognitive function. The maximum total score is 70 points, and the larger the score, the more severe the degree of impairment.
Time Frame: Baseline and 24 weeks
Population: Intent-to-treat (ITT) population. Last observation carried forward (LOCF) end point.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Group | Galantamine Group 1 | Galantamine Group 2
Number analyzed (Participants) | 191 | 191 | 192
Scores on a scale | 0.90 (5.89) | -0.58 (5.87) | -1.66 (5.37)
Statistical Analysis 1: Comparison: Placebo Group vs Galantamine Group 1; Test type: Superiority or Other; p = 0.0113, Least Square Means; Mean Difference (Final Values) = -1.49, 95% CI 2-sided [-2.64 to -0.34]
Statistical Analysis 2: Comparison: Placebo Group vs Galantamine Group 2; Test type: Superiority or Other; p < 0.0001, Least Square Means; Mean Difference (Final Values) = -2.59, 95% CI 2-sided [-3.74 to -1.44]

2. Primary Outcome: Distribution of Clinician's Interview-Based Impression of Change Plus - Japan (CIBIC Plus-J)
Description: CIBIC plus-J is the Japanese version of the Clinician's Interview-based Impression of Change plus the caregiver's input (CIBIC plus). It is a seven-point categorical assessment scale for evaluating the efficacy of antidementia drugs, ranging from "markedly improved" to "markedly worse".
Time Frame: 24 weeks
Population: Intent-to-treat (ITT) population. Last observation carried forward (LOCF) end point.
Measure: Number; unit: patients
Arm/Group | Placebo Group | Galantamine Group 1 | Galantamine Group 2
Number analyzed (Participants) | 191 | 191 | 192
patients
  Markedly improved | 0 | 0 | 1
  Moderately improved | 7 | 12 | 4
  Minimally improved | 36 | 39 | 32
  No change | 64 | 60 | 73
  Minimally worse | 62 | 64 | 61
  Moderately worse | 22 | 16 | 20
  Markedly worse | 0 | 0 | 1

3. Secondary Outcome: Change From Baseline in the Disability Assessment for Dementia (DAD)
Description: Each of the 40 item of the DAD is scored as 1 point= Yes, 0 point= No, or non applicable= N/A. A total score (minimum=0; maximum=40) is the sum of points for each questions converted out 100. Items rated as Not Applicable (N/A) are not considered for the total score. The final score is a percentage that gives an appreciation of global function in activity of daily life (ADL). Higher scores represent less disability in ADL while lower scores indicate more dysfunction.
Time Frame: Baseline and 24 weeks
Population: Intent-to-treat (ITT) population. Last observation carried forward (LOCF) end point.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Group | Galantamine Group 1 | Galantamine Group 2
Number analyzed (Participants) | 191 | 191 | 192
Scores on a scale | -2.8 (10.3) | -1.0 (9.4) | -2.2 (9.3)
Statistical Analysis 1: Comparison: Placebo Group vs Galantamine Group 1; Test type: Superiority or Other; p = 0.0774, Least Square Means; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-0.2 to 3.7]
Statistical Analysis 2: Comparison: Placebo Group vs Galantamine Group 2; Test type: Superiority or Other; p = 0.6207, Least Square Means; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.5 to 2.4]

4. Secondary Outcome: Change From Baseline in the Behavioral Pathology in Alzheimer's Disease Rating Scale (Behave-AD)
Description: Behave-AD is a CIBIC plus-J subscale that rates the patient's severity of psychotic symptoms. This four-point scale varies from 0 (=none) to 3 (= serious).
Time Frame: Baseline and 24 weeks
Population: Intent-to-treat (ITT) population. Last observation carried forward (LOCF) end point.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Group | Galantamine Group 1 | Galantamine Group 2
Number analyzed (Participants) | 191 | 191 | 192
Scores on a scale | 0.0 (3.1) | -0.2 (4.2) | -0.3 (3.1)
Statistical Analysis 1: Comparison: Placebo Group vs Galantamine Group 1; Test type: Superiority or Other; p = 0.8419, Least Square Means; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.6 to 0.8]
Statistical Analysis 2: Comparison: Placebo Group vs Galantamine Group 2; Test type: Superiority or Other; p = 0.7942, Least Square Means; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.8 to 0.6]

5. Secondary Outcome: Change From Baseline in the Mental Function Impairment Scale (MENFIS)
Description: MENFIS is a Clinician's Interview-Based Impression of Change (CIBIC) plus-Japan subscale that rates the patient's severity for mental function impairment. This seven-point scale varies from 0 (= absolutely no impairment) to 6 (=complete impairment).
Time Frame: Baseline and 24 weeks
Population: Intent-to-treat (ITT) population. Last observation carried forward (LOCF) end point.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Group | Galantamine Group 1 | Galantamine Group 2
Number analyzed (Participants) | 191 | 191 | 192
Scores on a scale | 2.2 (5.2) | 1.6 (5.2) | 1.9 (5.2)
Statistical Analysis 1: Comparison: Placebo Group vs Galantamine Group 1; Test type: Superiority or Other; p = 0.3141, Least Square Means; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.6 to 0.5]
Statistical Analysis 2: Comparison: Placebo Group vs Galantamine Group 2; Test type: Superiority or Other; p = 0.6089, Least Square Means; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.3 to 0.8]

ADVERSE EVENTS:
Time Frame: Approximately 28 weeks
Arm/Group | Placebo Group | Galantamine Group 1 | Galantamine Group 2
Serious Adverse Events (participants affected / at risk) | 13/194 | 7/192 | 8/194
Other Adverse Events (participants affected / at risk) | 146/194 | 154/192 | 163/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=194) | Galantamine Group 1 (N=192) | Galantamine Group 2 (N=194)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Anemia folate deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Respiration failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=194) | Galantamine Group 1 (N=192) | Galantamine Group 2 (N=194)
Nasopharyngitis (Infections and infestations) | 36 (57) | 40 (53) | 38 (51)
Anorexia (Metabolism and nutrition disorders) | 9 (12) | 18 (28) | 16 (20)
Decreased appetite (Metabolism and nutrition disorders) | 8 (11) | 10 (12) | 14 (18)
Headache (Nervous system disorders) | 17 (24) | 9 (10) | 11 (18)
Nausea (Gastrointestinal disorders) | 11 (15) | 24 (44) | 32 (61)
Vomiting (Gastrointestinal disorders) | 16 (20) | 26 (38) | 21 (44)
Diarrhoea (Gastrointestinal disorders) | 18 (23) | 19 (43) | 21 (31)
Constipation (Gastrointestinal disorders) | 4 (4) | 12 (13) | 6 (6)
Weight decreased (Investigations) | 5 (5) | 12 (12) | 10 (10)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 10 (10) | 10 (11)
Fall (Injury, poisoning and procedural complications) | 22 (28) | 22 (31) | 15 (18)
Contusion (Injury, poisoning and procedural complications) | 10 (11) | 10 (11) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the sponsor requires.